CLINICAL TRIAL: NCT01149226
Title: Effects of Chloral Hydrate on Induction, Maintenance, and Recovery From Sevoflurane Anesthesia in Day-case Pediatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Hae Keum Kil / Professor, Severance Hospital, YUHS
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2010-0084
Record Dates: First submitted 2010-06-16; First posted 2010-06-28 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Pediatric
Keywords: pediatric patients; ASA physical status I or II; aged between 1-5 yrs
MeSH Terms: interventions — Chloral Hydrate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo control (Placebo Comparator)
  Interventions: Drug: chloral hydrate
- oral medication chloral hydrate (Experimental)
  Interventions: Drug: chloral hydrate

INTERVENTIONS:
Drug: chloral hydrate — 30 min before the induction of anesthesia, chloral hydrate (40 mg/kg) or placebo was administered to the children orally.

SUMMARY:
Effects of Choral Hydrate on Induction, Maintenance, and Recovery from Sevoflurane Anesthesia in Day-case Pediatric Surgery

ELIGIBILITY:
Inclusion Criteria:

1. ASA I or II
2. 1-5 years children
3. elective day-case orchiopexy

Exclusion Criteria:

1. congenital hear disease
2. renal disease
3. liver disease
4. growth retardation
5. coagulopathy

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Preoperative Anxiety
  Preoperative Anxiety Score
  Modified Yale Preoperative Anxiety Scale (YPAS, 0-100) was assessed by observer Anesth Analg 1997;85:783-8
Induction Compliance
  Induction Compliance Checklist
  Induction Compliance Checklists (ICC, 0-10) was assessed by anesthetist Anesthesiology 1998;89:1147-56
Postoperative Pain
  -Postoperative Pain Score
  Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale (0-10) was assessed by observer Am J Crit Care. 2010 Jan;19(1):55-61
Posthospitalization Behavior
  Posthospitalization Behavior Questionnaire
  Posthospitalization Behavioural Questionnaire (27-135)was sent to all parents of children Paediatr Anaesth. 2001 Nov;11(6):719-23.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea